CLINICAL TRIAL: NCT03484507
Title: Parasitic Ulcer Treatment Trial Pilot
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Research to Prevent Blindness (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UCSF-IRB-17-23895
Record Dates: First submitted 2018-03-24; First posted 2018-03-30 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Acanthamoeba Keratitis
MeSH Terms: conditions — Acanthamoeba Keratitis | interventions — Chlorhexidine; Povidone-Iodine; prednisolone phosphate; Hypromellose Derivatives

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Chlorhexidine monotherapy (Active Comparator): Topical chlorhexidine 0.04%
  Interventions: Drug: Chlorhexidine
- Chlorhexidine plus povidone iodine (Experimental): Topical chlorhexidine 0.04% plus povidone iodine 2.5%
  Interventions: Drug: Chlorhexidine; Drug: Povidone-Iodine
- Early corticosteroids (Experimental): Topical prednisolone sodium phosophate 1% for weeks 4-11
  Interventions: Drug: Prednisolone Sodium Phosphate
- Late corticosteroids (Experimental): Artificial tears for weeks 4-5, then topical prednisolone sodium phosophate 1% for weeks 6-11
  Interventions: Drug: Prednisolone Sodium Phosphate; Drug: Hydroxypropyl Methylcellulose
- Placebo (Placebo Comparator): Artificial tears for weeks 4-11
  Interventions: Drug: Hydroxypropyl Methylcellulose

INTERVENTIONS:
Drug: Chlorhexidine — 1 drop half-hourly for days 1-2, then hourly for days 3-6, then 8 times daily until the 4-week visit
  Arms: Chlorhexidine monotherapy; Chlorhexidine plus povidone iodine
Drug: Povidone-Iodine — 1 drop half-hourly for days 1-2, then hourly for days 3-6, then 8 times daily until the 4-week visit
  Arms: Chlorhexidine plus povidone iodine
Drug: Prednisolone Sodium Phosphate — 1 drop 4 times daily for weeks 4-9, then 2 times daily for weeks 10-11
  Arms: Early corticosteroids
Drug: Hydroxypropyl Methylcellulose — 1 drop 4 times daily for weeks 4-9, then 2 times daily for weeks 10-11
  Arms: Placebo
Drug: Prednisolone Sodium Phosphate — 1 drop 4 times daily for weeks 6-9, then 2 times daily for weeks 10-11
  Arms: Late corticosteroids
Drug: Hydroxypropyl Methylcellulose — 1 drop 4 times daily for weeks 4-5
  Arms: Late corticosteroids

SUMMARY:
This is a study of optimal treatments for acanthamoeba keratitis. In the first part of the study, participants will be randomized to chlorhexidine monotherapy or chlorhexidine plus povidone iodine. After four weeks of therapy, participants will be re-randomized to early corticosteroids, later corticosteroids, or placebo.

DETAILED DESCRIPTION:
Acanthamoeba keratitis is a rare eye infection that is difficult to treat. The mainstay of therapy is a biguanide agent such as chlorhexidine, though recent studies have found povidone iodine to be effective for killing acanthamoeba organisms in vitro. Thus, we randomize participants to topical chlorhexidine 0.04% monotherapy (i.e., routine care) versus topical chlorhexidine 0.04% plus topical poviodine iodine 2.5%. The primary outcome is clearance of acanthamoeba from the ocular surface at 4 weeks.

The role of topical corticosteroids in acanthamoeba keratitis is controversial. Topical corticosteroids can promote growth of acanthamoeba, but may also reduce inflammation and vision-threatening complications of infection. Here, we randomize participants who have completed a course of anti-amoebic therapy to one of three groups: early prednisolone sodium phosphate 1% (started at 4 weeks), late prednisolone sodium phosphate 1% (started at 6 weeks) or placebo (started at 4 weeks). The primary outcome will be visual acuity at 6 months.

ELIGIBILITY:
Trial 1 Inclusion Criteria:

* Smear or culture positive for acanthamoeba
* Age 13 years or greater

Trial 1 Exclusion Criteria:

* Interstitial or viral keratitis on history or examination
* Corneal perforation
* Therapeutic keratoplasty for acanthamoeba keratitis
* Unwillingness or inability to follow-up (e.g., living too far from hospital)

Trial 2 Inclusion Criteria

* Smear or culture positive for acanthamoeba, with 4 weeks of anti-amoebic treatment
* Age 13 years or greater
* Willing to participate in study

Trial 2 Exclusion Criteria

* Interstitial or viral keratitis on history or examination
* Fungus identified on culture and smear after 2 weeks of anti-amoebic treatment
* Corneal perforation
* Therapeutic keratoplasty for acanthamoeba keratitis
* Unwillingness or inability to follow-up (e.g., living too far from hospital)

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Trial 1: Microbial clearance | 4 weeks
  Acanthamoeba culture
Trial 2: Best spectacle corrected visual acuity | 6 months

SECONDARY OUTCOMES:
Trial 1: Best spectacle corrected visual acuity | 4 weeks
Trial 1: Time to re-epithelialization | 4 weeks
Trial 1: Clinical cure | 4 weeks
Trial 2: Time to clinical cure | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy D Keenan, MD, Principal Investigator — University of California, San Francisco
Locations (2):
- India (2):
  - Aravind Eye Hospital, Coimbatore, Tamil Nadu
  - Aravind Eye Hospital, Madurai, Tamil Nadu

IPD SHARING:
Plan to Share IPD: No